CLINICAL TRIAL: NCT06451289
Title: Does Optic Nerve Sheath Diameter and Its Ratio to Eyeball Transverse Diameter Correlate With the Duration of Seizures in Post-ictal Children?
Brief Title: Study on Optic Nerve Sheath Diameter Measurements in Prolonged Pediatric Seizures
Acronym: ONSD
Status: Completed | Type: Observational
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, İpek Dokurel, Principal investigator, Balikesir University
Other Study IDs: ONSDseizureduration
Record Dates: First submitted 2024-06-03; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Intracranial Pressure Increase; Seizures; Children, Only
Keywords: Computed head tomography; Seizure; ONSD; elevated intracranial pressure
MeSH Terms: conditions — Intracranial Hypertension; Seizures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- postictal children: Postictal children aged one to 18 years who presented to the pediatric emergency department underwent head CT according to the Pediatric Emergency Care Applied Research Network (PECARN) guidelines. The seizures were observed by a health worker or directly with home videos.
  Interventions: Diagnostic Test: Head computered tomography
- the healthy controls: Previously healthy children admitted to the emergency department and having head CT without space-occupying/incidental lesions were determined as a control group.
  Interventions: Diagnostic Test: Head computered tomography

INTERVENTIONS:
Diagnostic Test: Head computered tomography — Retrospective data collecting from medical records

SUMMARY:
A total of 88 postictal children with generalized or focal seizures were included in the study.

The ONSD and ONSD/ETD ratio was measured independently by a pediatric neurologist and pediatric emergency expert, three times in both eyes using non-contrasted computed tomography taken within one hour after the seizure.

The characteristics of seizures (duration, etiology, initiated treatment, and frequency) were recorded.

Non-traumatic patients with normal head computed tomography findings at the hospital admission were considered as the control group (n=109).

DETAILED DESCRIPTION:
This was a prospective observational case-control study. The study included children aged 1 to 18 years who had undergone cranial CT scans in accordance with the Pediatric Emergency Care Applied Research Network (PECARN) guidelines between September 2020 and December 2022.

The seizures only observed by a health worker or directly with home videos were taken into consideration.

The definition of prolonged seizures proposed by the ILAE Task Force on Classification of Status Epilepticus was employed: those lasting more than five minutes for focal seizures and more than ten minutes for generalized seizures.

Children admitted to the emergency department and having head CT without space-occupying/incidental lesions were determined as a control group.

The participants were divided into two groups: postictal children (n=88) and healthy controls (n=109). Furthermore, the postictal children were divided into two groups, namely those with focal (n=56) and generalized (n=32) seizures.

The following variables were recorded from the medical records: patients' demographic characteristics (age, sex, body mass index), type of seizures (focal or generalized), the duration of seizures, seizure frequency, type of medication initiated, and the etiology of the seizures.

To ensure the highest standards of care, the pediatric head CTs were independently reviewed by a pediatric neurologist and a pediatric emergency expert.

The investigators measured Optic Nerve Sheath Diameter as a thickness at a distance of 3 mm from the optic disc.

The investigators measured the Eyeball Transverse Diameter via axial images, using the widest diameter of each eyeball from retina to retina.

The data were presented in the form of frequencies and percentiles for categorical variables and means with standard deviations (SDs) or medians with interquartile ranges for continuous variables.

The Mann-Whitney U tests were employed to ascertain the significance of the differences in ONSD and ONSD/ETD ratio observed between the independent groups.

A receiver operating curve (ROC) was constructed and the area under the curve (AUC) was measured in order to evaluate the discrimination ability.

ELIGIBILITY:
Inclusion Criteria:

* seizures were observed by a health worker or directly with home videos.
* prolonged seizures were used: those lasting more than 5 minutes for focal seizures and more than 10 minutes for generalized seizures.

Exclusion Criteria:

* Incomplete medical records; prior intracranial lesions, such as cysts (arachnoid, and pineal cysts),
* Chiari malformations, sequelae gliotic lesions, or incidental space-occupying lesions (cavernoma, lipoma, etc.);
* Chronic neuromuscular disease, metabolic or genetic disorders;
* Ocular trauma, periorbital cellulitis glaucoma, refraction errors, or optic disc drusen; or a history of retinopathy of prematurity
* Images with streak and movement artifacts, as well as images with pathologies that prevent measurement of the ONSD

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Postictal children with generalized or focal seizures were admitted to the emergency department after seizures and were taken non-contrasted computed head tomography within one hour after the seizure.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
elevated ICP in postictal cildren | 0-4 hours of emergengy department admission
  The investigators aim to show that elevated ICP which caused by prolonged seizures in children might be measured by optic nerve sheath diameter (ONSD) and ONSD/eyeball transverse diameter (ETD) ratios by head CT.
to prove seizures cause elevated ICP by measuring optic nerve sheath diameter (ONSD) and optic nerve in sheath diameter to eyeball transverse diameter (ETD) ratio and comparing these results with healthy controls | 4th to 5th hour of emergengy department admission
  The investigators aim to prove that pediatric seizures cause elevated ICP. This could be predicted by measuring optic nerve sheath diameter (ONSD) and optic nerve sheath diameter to eyeball transverse diameter (ETD) ratio. And compare these measurements with healthy controls.
to prove various seizure types cause variations in ICP and to show these can be detected by measuring optic nerve sheath diameter (ONSD) and optic nerve in sheath diameter to eyeball transverse diameter (ETD) ratio | 4th to 5th hour of emergengy department admission
  The investigators aim to detect the difference in ICP by measuring optic nerve sheath diameter (ONSD) and optic nerve sheath diameter to eyeball transverse diameter (ETD) ratio in children with focal and generalized seizures.And compare these results.

CONTACTS AND LOCATIONS:
Overall Officials: İpek Dokurel Çetin, MD, Principal Investigator — Balikesir Üniversity Medical faculty hospital
Locations (1):
- Balikesir Ataturk City Hospital, Balıkesir, Altieylul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Handan Gunsay R, Cikrikci Isik G, Yildirim M, Gokcek O, Korucu O, Cevik Y. Evaluation of postictal optic nerve sheath diameter at epileptic patients. Epilepsy Behav. 2023 Jul;144:109264. doi: 10.1016/j.yebeh.2023.109264. Epub 2023 May 27. PMID 37247582